CLINICAL TRIAL: NCT07283094
Title: FHD-286 With Low-Dose Weekly Decitabine/Venetoclax in Patients With Acute Myeloid Leukemia
Acronym: FHD-286
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Foghorn Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-16661; 2516661-FHD-286 (Other Grant/Funding Number: Foghorn Therapeutics)
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Decitabine; venetoclax

STUDY DESIGN:
Intervention Model Description: The study will enroll approximately 3-6 participants per cohort using a 3+3 design, resulting in a total of approximately 6-12 participants. During dose escalation, up to 5 additional participants per dose level may be enrolled at dose levels that have already been cleared. After a dose(s) has been selected for further study, additional participants may be enrolled to further explore safety or preliminary clinical activity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Decitabine, Venetoclax, and FHD-286 (Experimental): Administration:
  * Decitabine is reconstituted with 5 mL of sterile water and given by subcutaneous (SC) injection at the investigational site.
  * Venetoclax is taken as a tablet provided by the investigational site pharmacy or another authorized specialty pharmacy.
  * FHD-286 is taken as a capsule provided by the investigational site pharmacy.
  Interventions: Drug: Decitabine; Drug: Venetoclax; Drug: FHD-286

INTERVENTIONS:
Drug: Decitabine — Decitabine: 0.2 mg/kg/day subcutaneously once weekly (QW) (days 1, 8, 15, 22 [±3 days] of each 28-day cycle)
Drug: Venetoclax — Venetoclax: 400 mg orally (PO) (tablets) QW, concurrent with the first weekly DAC dose (days 1, 8, 15, and 22 [±1 day] of each 28-day cycle)
Drug: FHD-286 — FHD-286: 2.5 or 5 mg (based on the assigned dose group) PO (capsules) once daily (QD) 5 days per week (days 3-7, 10-14, 17-21, and 24-28 of each 28-day cycle).
  If acceptable safety and tolerability are observed at the end of cycle 1 with at least 3 DLT-evaluable participants in cohort 1 (FHD-286 2.5 mg QD), the dose of FHD-286 will be escalated to 5 mg QD for cohort 2

SUMMARY:
This is a Phase 1, uncontrolled, single-arm, open-label, nonrandomized, dose escalation, study of Decitabine (DAC)+Venetoclax (VEN)+FHD-286 in participants with newly diagnosed Acute Myeloid Leukemia (AML) classified as adverse risk per the 2022 European Leukemia Net (ELN) criteria or AML that has progressed after one prior line of therapy.

DETAILED DESCRIPTION:
This study evaluates the addition of FHD-286, which has a distinct mechanism of action and clinical activity in AML, to a modification of the current standard of care regimen (DAC/VEN) that has been shown to be more tolerable than and have similar clinical activity as the more intensive regimen evaluated in the VIALE-A study (see References section).

Total duration of trial intervention for each participant will vary. Participants are anticipated to remain on treatment for at least 12 weeks (induction period). As long as they are receiving benefit from treatment, participants may remain on treatment until they experience a reason for treatment discontinuation or study withdrawal. Participants may remain on study as long as they are receiving DAC and VEN, even if FHD-286 is on hold or discontinued due to toxicity.

After written informed consent is obtained from a participant, they will undergo screening evaluations within 28 days before the first dose of study treatment. Results from assessments conducted within 28 days before the first dose of study treatment may be used to fulfill screening requirements, even if they occurred before written informed consent was obtained. The first 3 to 6 participants will participate in the safety run-in portion of the study. During this portion, if ≥3 of the participants develop AEs meeting the stopping criterion during the DLT evaluation period, the study will be terminated. Thereafter, interim safety analyses will be conducted after the enrollment of every 3 participants. The first 12 weeks of treatment (cycles 1-3) are an induction period intended to produce a relatively rapid reduction in tumor burden, to a level that will permit more functional hematopoiesis, alleviating cytopenias and permitting bone marrow recovery. During the induction period, dose modifications and holds are discouraged, except in the case of severe toxicity from severe, non-hematologic adverse events. Additionally, if treatment-related myelosuppression is suspected, dose holds or reductions may be implemented, upon agreement with the principal investigator (PI). If the participant is receiving clinical benefit (at minimum, stable disease) after 12 weeks of treatment, they will have the option of continuing their treatment regimen during the long-term treatment period. The goal of the long-term treatment period is to continue to provide clinical benefit via disease control and hematopoietic improvement. Each participant may continue treatment until they experience a reason for treatment discontinuation. Upon discontinuation of treatment, each participant will be asked to undergo an end-of-treatment evaluation. Thirty days after discontinuation of study treatment, each participant will be asked to undergo a safety follow-up evaluation. Participants will then be contacted approximately every 2 months for long-term follow-up to assess survival status, receipt and type of subsequent anticancer therapy, and disease status.

Dose-limiting toxicities will be assessed during the first cycle (first 28 days) of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed adverse risk AML, including Myelodysplastic Syndrome/Acute Myeloid Leukemia (MDS/AML), per the 2022 ELN criteria, with a histopathologic diagnosis confirmed by hematopathology review OR AML that has progressed after 1 prior line of therapy
2. Aged ≥75 years, or aged 18-74 years and either refuse to receive intensive induction chemotherapy or are not a candidate for intensive induction chemotherapy due to one or more of the following comorbidities:

   1. Eastern Cooperative Oncology Group performance status (ECOG PS) of 2 or 3
   2. Cardiac history of congestive heart failure requiring treatment, ejection fraction ≤50%, or chronic stable angina pectoris
   3. Diffusing capacity of the lung for carbon monoxide ≤65% or forced expiratory volume in 1 second ≤65%
   4. Creatinine clearance ≥30 mL/min to <45 mL/min
   5. Moderate hepatic impairment with total bilirubin >1.5 to ≤3.0×upper limit of normal (ULN)
   6. Any other comorbidity that the investigator judges to be incompatible with intensive chemotherapy
3. Bone marrow blasts ≥10%
4. Have not received a hypomethylating agent (HMA) or VEN for their disease under study
5. No other disease-directed therapy, except hydroxyurea or cytarabine, and including experimental or investigational drug therapy, for at least 14 days before study entry
6. ECOG PS:

   1. ≥75 years: ≤2
   2. ≥18 years to <75 years: ≤3
7. Life expectancy ≥3 months
8. Adequate end organ function, defined as:

   1. Adequate hepatic function, including:

      * Serum total bilirubin ≤3.0×ULN, unless considered due to advanced hematologic malignancy involvement or documented Gilbert syndrome with direct bilirubin ≤1.5×ULN
      * Aspartate aminotransferase, alanine aminotransferase, and alkaline phosphatase ≤3.0×ULN, unless considered due to advanced hematologic malignancy involvement
   2. Prothrombin time ≤1.5×ULN or international normalized ratio ≤1.4
   3. Activated partial thromboplastin time ≤1.5×ULN Note: Individuals who have been receiving a stable dose of anticoagulation therapy without bleeding episodes for ≥12 weeks may be considered for the study
   4. No known portal vein thrombosis
   5. Glomerular filtration rate (GFR) ≥30 mL/min (based on a contemporary, widely accepted, and clinically applicable equation that estimates GFR or a measure of GFR)
9. Adequate cardiovascular, respiratory, and immune system function as evidenced by the below criterion and in the opinion of the investigator:

   a. Left ventricular ejection fraction (LVEF) of ≥40% by echocardiogram (ECHO)
10. White blood cell count ≤20×10^9/L (treatment with hydroxyurea or cytarabine ≤1 g/m2 to achieve this count is allowed before the start of study treatment and for up to 28 days after the start of study treatment)
11. Agree to abide by dietary and other considerations required during the study
12. Ability to understand and willingness to sign a written informed consent form and complete study-related procedures

Exclusion Criteria:

1. Acute promyelocytic leukemia
2. Core binding factor AML who is a candidate for intensive chemotherapy
3. Eligible for and willing to receive standard HMA/VEN therapy
4. Evidence (or suspicion) of extramedullary involvement
5. Prior treatment with azacitidine, DAC, VEN, or FHD-286
6. Currently pregnant or breast-feeding. Women of child-bearing potential (WOCBP) must have negative serum pregnancy test within 72 hours before treatment start. (NOTE: WOCBP is any biological female, regardless of sexual or gender orientation, having undergone tubal ligation, or remaining celibate by choice, who has not undergone a documented hysterectomy or bilateral oophorectomy or has had a menses any time in the preceding 12 months [therefore not naturally post-menopausal for >12 months].)
7. Planning to become pregnant within 1 year after start of study treatment
8. Uncontrolled intercurrent illness that could limit life expectancy or ability to complete study correlates. This includes, but is not limited to:

   1. Ongoing or active infection. Because patients with myeloid malignancies are prone to infections, if individuals are actively being treated with appropriate antibiotics or antifungal agents with clinical evidence of infection control, they may be considered for the study. If treatment with a triazole antifungal agent is indicated, isavuconazonium sulfate should be used preferentially. If isavuconazonium sulfate cannot be used, a different triazole antifungal agent may be used. Refer to Exclusion Criterion 10a regarding strong Cytochrome P450, family 3, subfamily A (CYP3A) inhibitors
   2. Uncontrolled concurrent malignancy
   3. Heart rate-corrected QT interval (QTc) by Fridericia method (QTcF) >470 milliseconds (ms) or other factors that increase the risk of QTc prolongation. Participants with QTcF >470 ms and bundle branch block and/or pacemaker rhythm may be considered for the study
   4. Congestive heart failure of New York Heart Association class III/IV. Individuals with compensated heart failure are permitted
   5. Unstable angina pectoris
   6. New or unstable cardiac arrhythmia. Patients with stable or controlled arrhythmias may be considered for the study.
   7. Decompensated liver cirrhosis (Child-Pugh score ≥12 or a Model for End-Stage Liver Disease (MELD) score ≥21)
   8. Psychiatric illness/social situation that would limit compliance with study requirements
   9. Any other prior or ongoing condition that, in the opinion of the investigator, could adversely affect the safety of the individual or impair the assessment of study results
9. Unable to tolerate administration of oral medication or has gastrointestinal dysfunction that would preclude adequate absorption, distribution, metabolism, or excretion of FHD-286.
10. Taking medications classified as:

    1. Strong CYP3A inhibitors. Individuals must have stopped treatment with strong CYP3A inhibitors at least 1 week or 5 half-lives, whichever is longer, before the first dose of study drug. Strong CYP3A inhibitors may be permitted; however, the FHD-286 dose should be reduced to 1.5 mg QD when a strong CYP3A inhibitor is in use, and for at least 1 week or 5 half-lives of the strong CYP3A inhibitor, whichever is longer, after the end of treatment with the strong CYP3A inhibitor. The venetoclax dose should be reduced as per the United States Prescribing Information (USPI)
    2. Strong CYP3A inducers. Individuals must have stopped treatment with strong CYP3A inducers at least 2 weeks or 5 half-lives, whichever is longer, before the first dose of study drug
    3. Sensitive CYP3A substrates with narrow therapeutic indices
11. Taking proton pump inhibitors (PPIs). Administration of PPIs must be stopped or switched to another acid-reducing agent (e.g., antacids or H2 blockers) at least 7 days before study entry
12. WOCBP sexually active with male partners and fertile males sexually active with WOCBP unwilling to agree to use dual contraceptive measures (i.e., hormonal or barrier method of birth control, abstinence, condom), beginning at the screening visit and continuing until 4 weeks after taking the last dose of DAC/VEN and 90 days after taking the last dose of FHD-286. Participants must agree to refrain from donating sperm/Ova from the screening visit through 90 days after the last dose of FHD-286
13. Uncontrolled active HIV infection, as this will further increase the risk for opportunistic infections. However, individuals with HIV with undetectable viral load by polymerase chain reaction, without opportunistic infection, with Cluster of Differentiation 4 count (CD4) count >200 cells/µL, and on a stable regimen of antiretroviral therapy would be eligible
14. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection, unless the individual has a sustained viral response to HCV treatment or immunity to prior HBV infection
15. Known allergy or hypersensitivity to any component of DAC, VEN, or FHD-286 formulations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) | Through the 12-week induction period
  Dose limiting toxicity is defined as any adverse event (AE) that occurs during the DLT evaluation period that also meets any one of the criteria for hematologic and non-hematologic AEs as defined by the protocol and determined by the Data and Safety Monitoring Committee (DSMC), with input from the clinical study team.
  All AEs that cannot clearly be determined to be unrelated to FHD-286 or the combination of FHD-286 with DAC and VEN will be considered relevant to determining DLTs and any other emergent toxicities that are not explicitly defined by the DLT criteria to determine if any warrant a DLT designation, including toxicities that begin after the DLT evaluation period will be reviewed by the DSMC with input from the clinical study team.
  The percentage of participants with DLTs will be summarized by cohort.
Frequency and severity of the adverse event of special interest (AESI) | Through the 12-week induction period
  Differentiation syndrome is an adverse event of special interest for FHD-286. Suspected or confirmed differentiation syndrome will be reported, at minimum, as an important medical event. All Grade ≥2 events of Differentiation syndrome will be reported. The percentage of participants with DLTs will be summarized by cohort.
Percentage of participants who are able to continue treatment | After 12-week induction period
  The percentage of participants who are able to continue treatment without dose interruptions, reductions, or delays during the 12-week induction period will be summarized. Dose interruptions and delays are defined as delaying or interrupting treatment due to toxicity or intolerability for >2 weeks.

SECONDARY OUTCOMES:
Hemoglobin (Hgb) laboratory level for safety assessments | Weekly during 12-week induction period
  Hemoglobin laboratory values outside of normal ranges defined as 12.2 - 15.3 g/dL. Hgb counts will be monitored as part of treatment response criteria. Values outside of normal ranges will be summarized.
Platelet (Plt) laboratory level for safety assessments | Weekly during 12-week induction period
  Platelet laboratory values outside of normal ranges defined as 150 - 400 thousands per microliter (k/uL). Along with other laboratory values, treatment-emergent decreases in platelet counts will be monitored as part of dose modification guidelines and elevated platelet counts will be monitored as part of differentiation syndrome criteria. Platelet counts will also be monitored as part of treatment response criteria. Values outside of normal ranges will be summarized.
Absolute Neutrophil Count (ANC) laboratory level for safety assessments | Weekly during 12-week induction period
  Absolute neutrophil count laboratory values outside of normal ranges defined as 1.80 - 7.70 k/uL. Along with other laboratory values, treatment-emergent decreases in ANC counts will be monitored as part of dose modification guidelines and elevated ANC counts will be monitored as part of differentiation syndrome criteria. ANC counts will also inform the need for supportive concomitant therapy. ANC counts will also be monitored as part of treatment response criteria. Values outside of normal ranges will be summarized.
Overall response rate (ORR) | End of Cycle 1 (28 days) and end of Cycle 2 (56 days)
  Overall response rate is defined as the rate of complete remission (CR), CR with incomplete hematologic recovery, morphologic leukemia-free state, and partial remission, based on ELN 2022 criteria. ORR will be summarized by cohort.
Duration of response | Up to 2 years
  Duration of response is defined as the time from the first documentation of a response until the first documentation of disease progression or relapse, or death.
Percentage of participants who achieve Complete Remission | End of Cycle 1 (28 days), end of Cycle 2 (56 days) and Cycle 3 (84 days)
  Complete remission is defined as bone marrow blasts <5%; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; ANC ≥1.0×10^9/L (1000/µL); platelet count ≥100×10^9/L (100,000/µL). The percentage of participants who achieve Complete Remission will be summarized by cohort and disease state.

CONTACTS AND LOCATIONS:
Overall Officials: Mendel R Goldfinger, MD, Principal Investigator — Montefiore Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dohner H, Wei AH, Appelbaum FR, Craddock C, DiNardo CD, Dombret H, Ebert BL, Fenaux P, Godley LA, Hasserjian RP, Larson RA, Levine RL, Miyazaki Y, Niederwieser D, Ossenkoppele G, Rollig C, Sierra J, Stein EM, Tallman MS, Tien HF, Wang J, Wierzbowska A, Lowenberg B. Diagnosis and management of AML in adults: 2022 recommendations from an international expert panel on behalf of the ELN. Blood. 2022 Sep 22;140(12):1345-1377. doi: 10.1182/blood.2022016867. PMID 35797463
- [Background] DiNardo CD, Jonas BA, Pullarkat V, Thirman MJ, Garcia JS, Wei AH, Konopleva M, Dohner H, Letai A, Fenaux P, Koller E, Havelange V, Leber B, Esteve J, Wang J, Pejsa V, Hajek R, Porkka K, Illes A, Lavie D, Lemoli RM, Yamamoto K, Yoon SS, Jang JH, Yeh SP, Turgut M, Hong WJ, Zhou Y, Potluri J, Pratz KW. Azacitidine and Venetoclax in Previously Untreated Acute Myeloid Leukemia. N Engl J Med. 2020 Aug 13;383(7):617-629. doi: 10.1056/NEJMoa2012971. PMID 32786187
- [Background] Aldoss I, Yang D, Aribi A, Ali H, Sandhu K, Al Malki MM, Mei M, Salhotra A, Khaled S, Nakamura R, Snyder D, O'Donnell M, Stein AS, Forman SJ, Marcucci G, Pullarkat V. Efficacy of the combination of venetoclax and hypomethylating agents in relapsed/refractory acute myeloid leukemia. Haematologica. 2018 Sep;103(9):e404-e407. doi: 10.3324/haematol.2018.188094. Epub 2018 Mar 15. No abstract available. PMID 29545346
- [Background] Pratz KW, Jonas BA, Pullarkat V, Thirman MJ, Garcia JS, Dohner H, Recher C, Fiedler W, Yamamoto K, Wang J, Yoon SS, Wolach O, Yeh SP, Leber B, Esteve J, Mayer J, Porkka K, Illes A, Lemoli RM, Turgut M, Ku G, Miller C, Zhou Y, Zhang M, Chyla B, Potluri J, DiNardo CD. Long-term follow-up of VIALE-A: Venetoclax and azacitidine in chemotherapy-ineligible untreated acute myeloid leukemia. Am J Hematol. 2024 Apr;99(4):615-624. doi: 10.1002/ajh.27246. Epub 2024 Feb 11. PMID 38343151
- [Background] Goldfinger M, Mantzaris I, Shastri A, Saunthararajah Y, Gritsman K, Sica RA, Kornblum N, Shah N, Levitz D, Rockwell B, Shapiro LC, Gupta R, Pradhan K, Xue X, Munoz A, Dhawan A, Fehn K, Comas M, Verceles JA, Jonas BA, Kambhampati S, Shi Y, Braunschweig I, Cooper DL, Konopleva M, Feldman EJ, Verma A. A weekly low-dose regimen of decitabine and venetoclax is efficacious and less myelotoxic in a racially diverse cohort. Blood. 2024 Nov 28;144(22):2360-2363. doi: 10.1182/blood.2024025834. PMID 39316768
- [Background] Velcheti V, Schrump D, Saunthararajah Y. Ultimate Precision: Targeting Cancer but Not Normal Self-replication. Am Soc Clin Oncol Educ Book. 2018 May 23;38:950-963. doi: 10.1200/EDBK_199753. PMID 30231326
- [Background] Saunthararajah Y, Sekeres M, Advani A, Mahfouz R, Durkin L, Radivoyevitch T, Englehaupt R, Juersivich J, Cooper K, Husseinzadeh H, Przychodzen B, Rump M, Hobson S, Earl M, Sobecks R, Dean R, Reu F, Tiu R, Hamilton B, Copelan E, Lichtin A, Hsi E, Kalaycio M, Maciejewski J. Evaluation of noncytotoxic DNMT1-depleting therapy in patients with myelodysplastic syndromes. J Clin Invest. 2015 Mar 2;125(3):1043-55. doi: 10.1172/JCI78789. Epub 2015 Jan 26. PMID 25621498
- [Background] Awada H, Mahfouz RZ, Kishtagari A, Kuzmanovic T, Durrani J, Kerr CM, Patel BJ, Visconte V, Radivoyevitch T, Lichtin A, Carraway HE, Maciejewski JP, Saunthararajah Y. Extended experience with a non-cytotoxic DNMT1-targeting regimen of decitabine to treat myeloid malignancies. Br J Haematol. 2020 Mar;188(6):924-929. doi: 10.1111/bjh.16281. Epub 2019 Nov 17. PMID 31736067
- [Background] Gu X, Tohme R, Tomlinson B, Sakre N, Hasipek M, Durkin L, Schuerger C, Grabowski D, Zidan AM, Radivoyevitch T, Hong C, Carraway H, Hamilton B, Sobecks R, Patel B, Jha BK, Hsi ED, Maciejewski J, Saunthararajah Y. Decitabine- and 5-azacytidine resistance emerges from adaptive responses of the pyrimidine metabolism network. Leukemia. 2021 Apr;35(4):1023-1036. doi: 10.1038/s41375-020-1003-x. Epub 2020 Aug 7. PMID 32770088
- [Background] Zavras PD, Shastri A, Goldfinger M, Verma AK, Saunthararajah Y. Clinical Trials Assessing Hypomethylating Agents Combined with Other Therapies: Causes for Failure and Potential Solutions. Clin Cancer Res. 2021 Dec 15;27(24):6653-6661. doi: 10.1158/1078-0432.CCR-21-2139. Epub 2021 Sep 22. PMID 34551907
- [Background] DiNardo CD, Fathi AT, Kishtagari A, Bhalla KN, Quintas-Cardama A, Reilly SA, Almon C, Patriquin C, Nabhan S, Healy K, Hickman D, Collins MP, Khalil A, Corrigan D, Zhao T, Piel J, Lyons K, Horrigan K, Schuck V, Martin P, Elliott G, Lahr DL, Bosinger M, D'Aco K, Smolen GA, Hentemann M, Loghavi S, Agresta S, Savona MR, Stein EM. A Phase I Study of FHD-286, a Dual BRG1/BRM (SMARCA4/SMARCA2) Inhibitor, in Patients with Advanced Myeloid Malignancies. Clin Cancer Res. 2025 Jun 13;31(12):2327-2338. doi: 10.1158/1078-0432.CCR-24-3790. PMID 40238563
- [Background] Jonas BA, Pollyea DA. How we use venetoclax with hypomethylating agents for the treatment of newly diagnosed patients with acute myeloid leukemia. Leukemia. 2019 Dec;33(12):2795-2804. doi: 10.1038/s41375-019-0612-8. Epub 2019 Oct 18. PMID 31628431
- [Background] Winters AC, Gutman JA, Purev E, Nakic M, Tobin J, Chase S, Kaiser J, Lyle L, Boggs C, Halsema K, Schowinsky JT, Rosser J, Ewalt MD, Siegele B, Rana V, Schuster S, Abbott D, Stevens BM, Jordan CT, Smith C, Pollyea DA. Real-world experience of venetoclax with azacitidine for untreated patients with acute myeloid leukemia. Blood Adv. 2019 Oct 22;3(20):2911-2919. doi: 10.1182/bloodadvances.2019000243. PMID 31648312
- [Background] Abaza Y, Winer ES, Murthy GSG, Shallis RM, Matthews AH, Badar T, Geramita EM, Kota VK, Swaroop A, Doukas P, Bradshaw D, Helenowski IB, Liu Y, Zhang H, Im A, Litzow MR, Perl AE, Atallah E, Altman JK. Clinical outcomes of hypomethylating agents plus Venetoclax as frontline treatment in patients 75 years and older with acute myeloid leukemia: Real-world data from eight US academic centers. Am J Hematol. 2024 Apr;99(4):606-614. doi: 10.1002/ajh.27231. Epub 2024 Feb 11. PMID 38342997
- [Background] Brandwein J, Page D, Liew E, Hnatiuk M, Bolster L, Hamilton M, Sawler D, Wang P. A Real-World Evaluation of Frontline Treatment for Acute Myeloid Leukemia With Azacitidine Plus Venetoclax. Clin Lymphoma Myeloma Leuk. 2025 Jul;25(7):e435-e442. doi: 10.1016/j.clml.2025.01.024. Epub 2025 Feb 1. PMID 40023757
- [Background] Short NJ, Daver N, Dinardo CD, Kadia T, Nasr LF, Macaron W, Yilmaz M, Borthakur G, Montalban-Bravo G, Garcia-Manero G, Issa GC, Chien KS, Jabbour E, Nasnas C, Huang X, Qiao W, Matthews J, Stojanik CJ, Patel KP, Abramova R, Thankachan J, Konopleva M, Kantarjian H, Ravandi F. Azacitidine, Venetoclax, and Gilteritinib in Newly Diagnosed and Relapsed or Refractory FLT3-Mutated AML. J Clin Oncol. 2024 May 1;42(13):1499-1508. doi: 10.1200/JCO.23.01911. Epub 2024 Jan 26. PMID 38277619
- [Background] DiNardo CD, Marvin-Peek J, Loghavi S, Takahashi K, Issa GC, Jen WY, Daver NG, Reville PK, Short NJ, Sasaki K, Mullin JK, Bradley CA, Borthakur G, Maiti A, Alvarado Y, Pemmaraju N, Abbas HA, Hammond DE, Haddad F, Bravo GM, Chien KS, Yilmaz M, Kornblau SM, Jabbour E, Ravandi F, Kadia T, Garcia-Manero G, Konopleva MY, Kantarjian HM. Outcomes of Frontline Triplet Regimens With a Hypomethylating Agent, Venetoclax, and Isocitrate Dehydrogenase Inhibitor for Intensive Chemotherapy-Ineligible Patients With Isocitrate Dehydrogenase-Mutated AML. J Clin Oncol. 2025 Aug 20;43(24):2692-2699. doi: 10.1200/JCO-25-00640. Epub 2025 Jun 13. PMID 40513054
- [Background] Fiskus W, Piel J, Collins M, Hentemann M, Cuglievan B, Mill CP, Birdwell CE, Das K, Davis JA, Hou H, Jain A, Malovannaya A, Kadia TM, Daver N, Sasaki K, Takahashi K, Hammond D, Reville PK, Wang J, Loghavi S, Sen R, Ruan X, Su X, Flores LB, DiNardo CD, Bhalla KN. BRG1/BRM inhibitor targets AML stem cells and exerts superior preclinical efficacy combined with BET or menin inhibitor. Blood. 2024 May 16;143(20):2059-2072. doi: 10.1182/blood.2023022832. PMID 38437498
- [Background] DiNardo CD, Roboz GJ, Watts JM, Madanat YF, Prince GT, Baratam P, de Botton S, Stein A, Foran JM, Arellano ML, Sallman DA, Hossain M, Marchione DM, Bai X, Patel PA, Kapsalis SM, Garcia-Manero G, Fathi AT. Final phase 1 substudy results of ivosidenib for patients with mutant IDH1 relapsed/refractory myelodysplastic syndrome. Blood Adv. 2024 Aug 13;8(15):4209-4220. doi: 10.1182/bloodadvances.2023012302. PMID 38640348
- [Background] Lee SH, Erber WN, Porwit A, Tomonaga M, Peterson LC; International Council for Standardization In Hematology. ICSH guidelines for the standardization of bone marrow specimens and reports. Int J Lab Hematol. 2008 Oct;30(5):349-64. doi: 10.1111/j.1751-553X.2008.01100.x. PMID 18822060
- [Background] Norsworthy KJ, Mulkey F, Scott EC, Ward AF, Przepiorka D, Charlab R, Dorff SE, Deisseroth A, Kazandjian D, Sridhara R, Beaver JA, Farrell AT, de Claro RA, Pazdur R. Differentiation Syndrome with Ivosidenib and Enasidenib Treatment in Patients with Relapsed or Refractory IDH-Mutated AML: A U.S. Food and Drug Administration Systematic Analysis. Clin Cancer Res. 2020 Aug 15;26(16):4280-4288. doi: 10.1158/1078-0432.CCR-20-0834. Epub 2020 May 11. PMID 32393603
- [Background] Montesinos P, Bergua JM, Vellenga E, Rayon C, Parody R, de la Serna J, Leon A, Esteve J, Milone G, Deben G, Rivas C, Gonzalez M, Tormo M, Diaz-Mediavilla J, Gonzalez JD, Negri S, Amutio E, Brunet S, Lowenberg B, Sanz MA. Differentiation syndrome in patients with acute promyelocytic leukemia treated with all-trans retinoic acid and anthracycline chemotherapy: characteristics, outcome, and prognostic factors. Blood. 2009 Jan 22;113(4):775-83. doi: 10.1182/blood-2008-07-168617. Epub 2008 Oct 22. PMID 18945964
- [Background] Stahl M, Tallman MS. Differentiation syndrome in acute promyelocytic leukaemia. Br J Haematol. 2019 Oct;187(2):157-162. doi: 10.1111/bjh.16151. Epub 2019 Aug 13. PMID 31410848
- [Background] Gu X, Tohme R, Goldfinger M, et al: Venetoclax inhibition of pyrimidine synthesis guides methods for integration with decitabine or 5-azacytidine that are non-myelosuppressive. Presented at the 62nd ASH Annual Meeting and Exposition, Virtual, 05-08 Dec, 2020
- [Background] Dinardo CD, Kishtagari A, Ball B, et al: Preliminary safety, pharmacokinetic, and clinical activity results with FHD-286, a BRG1/BRM inhibitor, plus decitabine in a Phase 1 study in patients with relapsed or refractory myeloid malignancies. Presented at the EHA2025 Congress, Milan, Italy, 12-15 Jun, 2025
- [Background] Fiskus W, Piel J, Hentemann M, et al: Pre-clinical efficacy of targeting BAF complexes through inhibition of the dual ATPases BRG1 and BRM by FHD-286 in cellular models of AML of diverse genetic background. Presented at the American Society of Hematology (ASH) Annual Meeting & Exposition, New Orleans, Louisiana, 10-13 December, 2022
- [Background] Ueda M, El-Jurdi N, Cooper B, Caimi P, Baer L, Kolk M, Brister L, Wald DN, Otegbeye F, Lazarus HM, Sandmaier BM, William B, Saunthararajah Y, Woost P, Jacobberger JW, de Lima M. Low-Dose Azacitidine with DNMT1 Level Monitoring to Treat Post-Transplantation Acute Myelogenous Leukemia or Myelodysplastic Syndrome Relapse. Biol Blood Marrow Transplant. 2019 Jun;25(6):1122-1127. doi: 10.1016/j.bbmt.2018.12.764. Epub 2018 Dec 30. PMID 30599207